CLINICAL TRIAL: NCT04134312
Title: A Phase 1 Open Label Trial of Intravenous Administration of MVA-BN-Brachyury Vaccine in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVA-BN-BRACHY-IV-001
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Solid Metastatic Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MVA-BN-Brachyury IV (Experimental): MVA-BN-Brachyury will be administered intravenously every three weeks with three administrations in total at the dose indicated by the enrolled cohort.
  Interventions: Biological: MVA-BN-Brachyury

INTERVENTIONS:
Biological: MVA-BN-Brachyury — MVA-BN-Brachyury will be administered intravenously every three weeks with three administrations in total at the dose indicated by the enrolled cohort.

SUMMARY:
A Phase 1 open label trial of intravenous administration of MVA-BN-Brachyury vaccine in patients with advanced cancer. Patients with metastatic or unresectable locally advanced malignant solid tumors will be enrolled and treated according to a 3+3 dose escalation scheme. Up to 3 dose levels will be explored. Patients will receive MVA-BN-Brachyury every three weeks, three administrations in total. Patients will be hospitalized after each vaccination, over 48 hours. Trial duration will be approximately 24 weeks per patient including 3 months after the last vaccination follow up (FU) period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women > 18 years old.
2. Patients must be able to understand and be willing to sign a written informed consent document.
3. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
4. Eligible patients must have one of the histologically confirmed cancers and treatment history as described:

   * Chordoma

     * Symptomatic, unresectable, locally recurrent, or metastatic tumors are acceptable for enrollment, given that this represents incurable disease.
     * Only curative interventions are required as prior therapy (surgery or definitive radiation) as no known systemic therapies have proven benefit.
   * Non-Small Cell Lung Cancer

     * Metastatic or incurable locally advanced.
     * Disease progression after indicated targeted therapy (EGFR-mut, ALK-fusion, BRAF-mut).
     * Disease progression after one regimen of chemotherapy and anti-PD-1/L1 therapy either sequentially or concurrently.
   * Small Cell Lung Cancer

     * Metastatic disease.
     * Disease progression after 1st line chemotherapy.
   * Breast

     * Metastatic disease considered to be incurable.
     * Triple negative - disease progression after first line chemotherapy.
     * ER+ disease - must have had disease progression through at least 2 lines of hormonal therapy and at least 1 chemotherapy regimen.
     * Her2+ disease - must have had disease progression after at least 2 Her2-targeted therapy containing regimens.
     * ER+ and Her2+ - must meet requirements of each tumor marker subtype (see above).
   * Ovarian

     * Metastatic disease.
     * Disease progression after treatment with platinum-based chemotherapy.
   * Prostate

     * Metastatic Castration Resistant Prostate Cancer (mCRPC) AND
     * Disease progression after at least one line of treatment of abiraterone or enzalutamide and docetaxel.
   * Colorectal

     * Metastatic disease.
     * Must have received chemotherapy regimens containing 5-FU, oxaliplatin, irinotecan, and EGFR-targeted antibodies when indicated (absence of RAS mutation) with evidence of disease progression or AEs that preclude further treatment with standard therapies.
   * Pancreatic

     * Metastatic disease.
     * Disease progression after or intolerance to standard chemotherapy regimens of known benefit (FOLFIRINOX or Gemcitabine and Abraxane).
   * Hepatocellular

     * Incurable disease: liver only or metastatic.
     * Disease progression after at least one systemic therapy of known benefit (e.g. sorafenib).
   * Bladder

     * Metastatic disease.
     * At least one line of chemotherapy and immune checkpoint inhibitors second line.
   * Kidney

     * Metastatic disease.
     * After VEGF inhibitors, immune check-point inhibitors, m-TOR inhibitors.
5. Patients must have measurable or evaluable disease. Measurable disease is defined by RECIST 1.1. In the case of evaluable disease, patients should have cancer-related symptoms to justify risk.

   Evaluable disease is defined as any of the following:
   * Elevated serum tumor marker known to be related to the patient's tumor.
   * Clear radiographic or physical exam evidence of tumor which does not meet RECIST 1.1 measurement requirements.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Patients must have normal organ and bone marrow function as defined below:

   Renal function:
   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):
   * Female CrCl = [(140 - age in years) x weight in kg x 0.85] / [72 x serum creatinine in mg/dL]
   * Male CrCl = [(140 - age in years) x weight in kg x 1.00] / [72 x serum creatinine in mg/dL]

   Liver function:
   * Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3 x the ULN.
   * Total bilirubin ≤ 1.5 x ULN (in subjects with Gilbert's syndrome a total bilirubin ≤ 3.0 x ULN), or < 5 x ULN, if liver metastases are present.

   Hematological parameters (within one week of starting therapy):
   * Hemoglobin > 9 g/dL.
   * Platelet count ≥ 100,000/µL.
   * Absolute neutrophil count (ANC) ≥ 1/ µL.
8. Troponin I within normal limits.
9. Electrocardiogram (ECG) without clinically significant findings.
10. Any prior chemotherapy, immunotherapy and/or radiation must be completed at least 4 weeks prior to the first planned dose of MVA-BN-Brachyury vaccine, with the following exceptions, assuming any toxicity related to these therapies is well controlled or resolved and the patient has been on that therapy for at least 8 weeks at the time of enrollment:

    * Prostate cancer - patients must continue to receive Gonadotropin-Releasing-Hormone (GnRH) agonist or antagonist therapy (unless orchiectomy has been done). Patients on abiraterone or enzalutamide may continue those therapies.
    * Breast cancer - patients may remain on hormonal therapy if indicated (Estrogen Receptor/Progesterone Receptor positive [ER/PR+]).
11. A minimum of 6 weeks from any prior antibody therapies (such as ipilimumab or anti-Programmed Death 1/Programmed Death Ligand 1[PD1/PD-L1]) is required due to prolonged half-life.
12. Patients must have recovered (grade 1 or baseline) from any clinically significant toxicity associated with prior therapy.
13. Women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test within 48 hours prior to administration of MVA-BN-Brachyury vaccine. Both men and women must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) through the trial treatment period and for at least three months after the last vaccination with MVA-BN-Brachyury vaccine.

Exclusion Criteria:

1. Receipt of an investigational agent within 28 days of the first planned dose of MVA-BN-Brachyury vaccine.
2. Concurrent chemotherapy or radiotherapy or other immunotherapy not explicitly allowed by inclusion criteria for this trial.
3. Known metastatic disease to the central nervous system, unless previously treated and well controlled for at least 3 months (clinically stable, no edema, no steroid treatment required).
4. History of anaphylaxis or severe allergic reaction to any vaccine, aminoglycoside antibiotics or egg products.
5. Active infection within 72 hours prior to vaccination.
6. Administration of antibiotics within 7 days prior to initial vaccination.
7. Subjects having known evidence of being immunocompromised as listed below:

   * Human immunodeficiency virus (HIV) positivity, active chronic hepatitis infection, including B and C.
   * Active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, and psoriasis not requiring systemic treatment are permitted.
   * Immunosuppressive therapy for post-organ transplant.
   * Chronic administration (defined as > 5 consecutive days of > 15 mg of prednisone (or equivalent) per day) of systemic corticosteroids within 14 days of the first planned dose of MVA-BN-Brachyury vaccine. Use of inhaled steroids, nasal sprays, eye drops, and topical creams is allowed. Steroids premedication for CT scans is allowed.
8. Vaccinations or planned vaccinations with a live vaccine within 30 days prior to the trial vaccination or with an inactivated vaccine within 14 days prior to the trial vaccination.
9. Patients with history of myocardial infarction, unstable angina pectoris, history of or existing CHF (NYHA Class II -IV), other cardiomyopathy, cardiac arrhythmia requiring medical treatment, clinically significant cardiac valvular disease, poorly controlled hypertension and hemodynamic effective pericardial effusion.
10. Known history of, or any evidence of active, non-infectious pneumonitis or primary pulmonary fibrosis.
11. Psychiatric illness/social situations that, in the opinion of the Investigator, would limit compliance with trial requirements.
12. Pregnant or breastfeeding women.
13. Any other condition, which in the opinion of the Investigator, would indicate the subject is a poor candidate for treatment with MVA-BN-Brachyury vaccine or would interfere with the evaluation of the trial endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Patients with Dose Limiting Toxicity (DLT) | DLT assessment is done 7 days after 2nd vaccination of last patient in each dose level
  Frequency of patients with DLTs

CONTACTS AND LOCATIONS:
Overall Officials: Marijo Bilusic, MD,PhD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeMaria PJ, Lee-Wisdom K, Donahue RN, Madan RA, Karzai F, Schwab A, Palena C, Jochems C, Floudas C, Strauss J, Marte JL, Redman JM, Dombi E, Widemann B, Korchin B, Adams T, Pico-Navarro C, Heery C, Schlom J, Gulley JL, Bilusic M. Phase 1 open-label trial of intravenous administration of MVA-BN-brachyury-TRICOM vaccine in patients with advanced cancer. J Immunother Cancer. 2021 Sep;9(9):e003238. doi: 10.1136/jitc-2021-003238. PMID 34479925
- [Derived] Wedekind MF, Widemann BC, Cote G. Chordoma: Current status, problems, and future directions. Curr Probl Cancer. 2021 Aug;45(4):100771. doi: 10.1016/j.currproblcancer.2021.100771. Epub 2021 Jul 1. PMID 34266694